CLINICAL TRIAL: NCT05724238
Title: The Effects of Traditional Herbal Dietary Supplements on General Fatigue and Negative Emotions of Graduate Students: A Randomized, Placebo-controlled Study
Brief Title: The Effects of Traditional Herbal Dietary Supplements on General Fatigue and Negative Emotions of Graduate Students
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Hsin-Jen Chen, Associate Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YM109050F
Record Dates: First submitted 2023-01-19; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Fatigue
Keywords: Astragalus; Traditional Herb; Fatigue; Negative Emotions; Graduate Students; Young Researchers
MeSH Terms: conditions — Fatigue

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Herbal Supplements (Experimental): Traditional Herbal Supplements (Kuan Sin Yin)
  Interventions: Dietary Supplement: Traditional Herbal Supplements (Kuan Sin Yin)
- Placebo (Placebo Comparator): Placebo starch powder with 10% Kuan Sin Yin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Traditional Herbal Supplements (Kuan Sin Yin) — Astragalus-based Kuan Sin Yin
  Arms: Traditional Herbal Supplements
Dietary Supplement: Placebo — Placebo starch powder with 10% Kuan Sin Yin
  Arms: Placebo

SUMMARY:
The goal of this randomized controlled trial is to determine the effect of traditional herbal supplements on general fatigue and negative emotions in generally healthy graduate students. The main questions it aims to answer are:

• Whether the traditional herbal supplements can ameliorate fatigue and negative emotions of young adults

DETAILED DESCRIPTION:
Participants will:

* Take oral herbal supplements or placebo as randomized for four weeks
* Be evaluated for the fatigue, anxiety, and depression levels at baseline and four weeks after the intervention
* Record sleep variables each day for five weeks

Researchers will compare the intervention group (receiving herbal supplements) with the placebo group (receiving placebo) to see if oral herbal supplements have effects on the outcomes and to examine the anti-fatigue effect two weeks after intervention.

ELIGIBILITY:
Inclusion Criteria:

* Scoring at least 4 points on the dichotomous Chalder's Fatigue Scale at baseline
* Working on at least one ongoing research project and expecting to continue working for at least one month

Exclusion Criteria:

* Taking medications as:
* Antidepressants
* Anxiolytics
* CNS stimulants
* Immunosuppressants
* With underlying diseases as:
* Diabetes mellitus
* Hematologic diseases
* Other major diseases as defined my MOHW of Taiwan

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Fatigue Level to Four Weeks | At week one (baseline) and week five (four weeks after the intervention)
  Measured by validated Chinese version of Chalder's Fatigue Scale, the score of which ranges from 0-33, with the higher representing a higher fatigue level (i.e. a worse outcome).

SECONDARY OUTCOMES:
Change from Baseline Sleep Quality to Four Weeks | At week one and week five
  Measured by the Chinese version of PSQI (Pittsburgh Sleep Quality Index), the score of which ranges from 0-21, with the higher representing a worse sleep quality (i.e. a worse outcome).
Change from Baseline Negative Emotion Scores to Four Weeks | At week one and week five
  Measured by the Chinese version of DASS-21 (Depression, Anxiety and Stress Scale-21 Items), the score of which ranges from 0-63, with the higher scores representing a higher negative emotion level (i.e. a worse outcome).
Change from Baseline Negative Emotion States to Four Weeks | At week one and week five
  Measured by the Chinese version of STAI-Y (State Trait Anxiety Inventory-Form Y), the score of which ranges from 20-80, with the higher representing a higher negative emotion level (i.e. a worse outcome).
Sleep Variables (Efficiency, Length, Midsleep time) | Each day from week one through week five
  Measured by sleep diary
Change from Baseline Fatigue At Each Week up to Six Weeks | Each week since week one until week seven
  Measured by validated Chinese version of Chalder's Fatigue Scale, the score of which ranges from 0-33, with the higher representing a higher fatigue level (i.e. a worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Hsin-Jen Chen, PhD, Principal Investigator — National Yang Ming Chiao Tung University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No